CLINICAL TRIAL: NCT06324422
Title: Can High-intensity Exercise be Used to Treat Fatigue in Parkinson´s Disease?
Brief Title: Exercise as Treatment of Fatigue in Parkinson´s Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fatigue & Parkinson's disease
Record Dates: First submitted 2024-03-07; First posted 2024-03-22 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease
Keywords: Exercise therapy; Parkinson's disease; Rehabilitation; Aerobic exercise; Resistance exercise; Fatigue
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized controlled multi-site trial with follow-up
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental): Participants must be clinically fatigued when enrolled and furthermore meet additional inclusion criteria.
  Interventions: Other: Aerobic exercise intervention
- Waitlist control group/resistance exercise group (Experimental): Participants must be clinically fatigued when enrolled and furthermore meet additional inclusion criteria.
  Interventions: Other: Resistance exercise intervention

INTERVENTIONS:
Other: Aerobic exercise intervention — Participants in this arm are randomized to perform 12 weeks of supervised high intensity progressive aerobic exercise comprising continuous and/or interval cycling-, rowing- or cross-trainer sessions, increasing from 30 minutes towards 60 minutes with intensity increasing from 65 to 90% of individual maximum heart rate. The 12 weeks of aerobic exercise are followed by 12 weeks of habitual lifestyle (follow up period).
  Arms: Aerobic exercise group
Other: Resistance exercise intervention — Participants in this arm are randomized to a 24-week waitlist control group. The control group will continue their habitual lifestyle throughout the 24 weeks. After 24 weeks, the waitlist control group will begin a 12 week supervised resistance exercise intervention comprising machine exercises in 3 to 5 sets with 2-3 minutes rest in between and a decrease from 12 to 6 repetitions in parallel with intensity increasing from 15RM (repetition maximum) to 8 RM.
  Arms: Waitlist control group/resistance exercise group

SUMMARY:
The primary goal of this study is to test whether 12 weeks of high-intensity aerobic exercise can treat fatigue in Parkinsons disease (PD).

The study will be a randomized multi-site controlled trial with follow up. Clinically fatigued persons with PD will be allocated to either 12 weeks of high-intensity aerobic exercise or to a waitlist control group receiving high-intensity resistance exercise after 24 weeks of habitual lifestyle (control period).

It is hypothesized that persons with PD receiving 12 weeks of high-intensity aerobic exercise will show superior effects on perceived fatigue (i.e., clinical relevant reductions) when compared to the PD control group (primary hypothesis), and that these effects are sustained after 12-weeks of follow up (secondary hypothesis).

DETAILED DESCRIPTION:
Background:

Parkinson's disease (PD) is a neurodegenerative disorder characterized by progressive and disabling motor and non-motor symptoms. Worldwide, PD is the fastest growing neurological disorder. Medical and surgical approaches in the symptomatic treatment of PD are progressing, but currently no disease modifying therapies exist. While awaiting effective disease modifying therapies, there is a major need to optimise symptomatic treatments of disabling PD symptoms.

A recent survey among 678 persons with PD (pwPD) and 104 carer/partner/family members or friends identified "Fatigue and energy" as the non-motor symptom that, if improved, would make the most marked difference to their daily lives. Fatigue affects 30-70% (depending on definition) of pwPD, and has been associated with worse prognosis, depression, anxiety, poor sleep, limited working ability, social distancing, decreased physical activity and impaired quality of life. Nevertheless, no effective medical or non-medical treatments exist for fatigue in PD.

Generally, physical exercise is highly recommended as a symptomatic intervention in PD. In a recent survey, 19% of pwPD (n=195) reported exercise as a coping strategy for fatigue and approximately half of the participants (49.7%, n=511) reported that exercise improved fatigue. However, it was not specified whether exercise was used as an acute coping strategy that instantly reduced/prevented fatigue, or if it was used as a chronic coping strategy, where regular exercise sessions reduced the chronic fatigue level. In other populations a physical exercise session can acutely lower the perceived fatigue level, while increasing the perceived energy level. To our knowledge, no studies have so far investigated the acute effects of different types of high intensity exercise on fatigue in pwPD.

Diverging evidence exists on the effects of regular exercise on fatigue in PD. Two thirds of the existing studies cautiously suggest that exercise (i.e., dance, aerobic exercise, exergaming, and mixed modalities) can potentially improve perceived fatigue. However, the last third show no difference or even increased fatigue levels following an exercise intervention. These heterogeneous results may be due to poor study designs as only one study applied fatigue as the primary outcome making most existing studies at risk of being underpowered. Also, none of the studies applied "clinical fatigue" as an inclusion criterium, which might have led to an underestimation of the potential exercise effects. Lastly, most existing studies were based on small sample sizes (i.e., <30 participants), half included no control group and most interventions prescribed exercise with low to moderate intensity (rather than higher intensity exercise), potentially limiting the effects of the intervention. Consequently, there is a need for a new PD high intensity exercise study with stronger methodologies assessing the chronic effects on fatigue.

Another argument for further evaluation of exercise as a treatment for fatigue in pwPD is based on findings from other neurological disorders such as multiple sclerosis, where both aerobic- and resistance exercise effectively reduce self-reported fatigue. Nonetheless, it remains unclear whether some exercise modalities are more efficient than others at inducing acute and chronic effects, making aerobic- and resistance exercise relevant for testing in pwPD.

Taken together, there is a need to investigate if high-intensity exercise can decrease fatigue in clinically fatigued pwPD, both acutely (i.e., effects observed immediately after a single exercise session) and/or chronically (i.e., the general fatigue level after a period with regular exercise sessions). Understanding the efficacy of basic exercise modalities (i.e., aerobic- and resistance exercise) and their working mechanisms before applying mixed exercise modalities therefore seems essential in the development of new fatigue management interventions for pwPD.

To gain further insight into the effects of high-intensity exercise on fatigue in PD, a randomized controlled multi-site trial with a follow up was designed.

As the present study may pave the way for introducing exercise in the management of PD fatigue, the study poses the potential to change clinical practice for pwPD.

The purpose of the mother study is to test the hypotheses that clinically fatigued pwPD receiving aerobic exercise will show superior effects on fatigue (i.e., clinical relevant reductions) when compared to a control group (primary hypothesis), and that these effects are sustained after 12 weeks of follow up (secondary hypothesis).

Interventions:

Aerobic exercise: 12 weeks, with 2-3 sessions per week, of supervised high intensity progressive aerobic exercise are performed comprising continuous and/or interval cycling-, rowing- or cross-trainer sessions, increasing from 30 towards 60 min with intensity increasing from 65 to 90% of individual maximum heart rate.

Resistance exercise: 12 weeks, with 2-3 sessions per week, of supervised resistance exercise are performed comprising machine exercises in 3 to 5 sets with 2-3 minutes rest in between and a decrease from 12 to 6 repetitions in parallel with intensity increasing from 15RM (repetition maximum) to 8 RM.

The exercise interventions have previously been used by our research group in neurological populations and are safe and feasible. Interventions are allowed to run up to 14 weeks to catch up missing exercise sessions.

Outcomes:

See the section "Outcome Measures" for specifications. Additionally, contact information, demographic information, health and medication information, and a blood sample will be obtained

Statistical considerations:

Whilst fatigue has been reported to decrease in pwPD after exercise interventions, none of the existing studies have applied the Modified Fatigue Impact Scale (MFIS). In fatigued persons with multiple sclerosis (MFIS ≥38 points) our group has previously shown that the total MFIS score can be substantially reduced following aerobic exercise (change scores: exercise -13±16 vs. control -3±16)28. By expecting comparable effects in fatigued pwPD, our sample size estimation (alpha level 5%, beta level 80%) revealed that a minimum of 84 pwPD must be enrolled in the study (i.e., n=42 for the aerobic exercise group and n=42 for the control group/waitlist resistance exercise group). Assuming a dropout of 10%, n=47 participants are required in each group.

Randomization:

After baseline assessment of fatigued participants, participants will be randomized in a 1:1 ratio to aerobic exercise or a waitlist control group. A computer-generated list of random numbers will be generated in the Research Electronic Data Capture (REDCap) system. The randomization will be stratified by site. The outcome assessors will be blinded for the randomization.

Perspectives:

The findings of this project hold the potential to establish aerobic exercise and/or resistance exercise as a safe and accessible treatment(s) of a frequent and disabling PD non-motor symptom, namely fatigue. In addition, the proposed study will expand our current knowledge about the acute effects of exercise on fatigue, potentially offering a simple modality to manage fatigue during everyday life. Taken together, the present study may lay the ground for a yet unexplored area of research with important implications for millions of pwPD, clinicians and the society.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 40 years
* Diagnosed with Idiopathic Parkinsons disease
* Stable in medical treatment for six month
* Able to transport themselves to and from exercise and testing sessions (with or without assistance)
* H&Y score of three or lower

Exclusion criteria:

* Performing high-intensity exercise more than two times per week
* Significant medical comorbidities such as cardiovascular, respiratory, orthopedic, metabolic, or other neurological disorders
* Cognitive dysfunction that prevents following or understanding instructions related to training and testing (answering questionnaires)
* Known depression or alcohol abuse

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Fatigue Impact Scale | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  Questionnaire assessing the effects of fatigue on physical, cognitive and psychosocial functioning. The total score of the MFIS is the sum of the scores for the 21 items and ranges from 0 to 84. The ranges of scores for each subscale are as follows: physical, 0 to 36; cognitive, 0 to 40; and psychosocial, 0 to 8. A higher score represents a higher impact of fatigue, in general or in relation to one of the above mentioned areas

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  A 9-item questionnaire which measures the severity of fatigue and its effect on patients activities and lifestyle. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score is 9 and maximum score possible is 63. Higher the score means greater fatigue severity.
Change in Parkinson's Fatigue Scale | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Parkinson Fatigue Scale is a 16-item patient rated scale that reflects the physical aspects of fatigue in patients with Parkinson's Disease and measures both the presence of fatigue and its impact on daily function. A total score is ranging from 16-80.
Change in Parkinson's Disease Questionnaire 39 | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Parkinson's Disease Questionnaire 39 is a tool used to assess the quality of life in individuals with Parkinson's disease. It consists of 39 questions across eight domains related to daily functioning and well-being. Each question is scored from 0 to 4, with higher scores indicating greater impairment. A lower total score suggests a better quality of life, while higher scores indicate poorer quality of life. The total score ranges from 0 to 156.
Change in Baecke Habitual Physical Activity Questionnaire | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Baecke Habitual Physical Activity Questionnaire is a tool used to assess an individual's level of physical activity in their daily life. It consists of a series of questions covering three domains: work-related physical activity, sports-related physical activity, and leisure-time physical activity. Each domain assesses the frequency, intensity, and duration of physical activities performed by the individual. The questionnaire aims to capture the overall level of physical activity and its distribution across different life domains. Higher scores indicate a higher level of physical activity.
Change in Pitchburg Sleep Quality Index | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Pittsburgh Sleep Quality Index is a questionnaire used to assess sleep quality over a one-month time interval. It comprises 19 items covering seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored on a scale from 0 to 3, with higher scores indicating poorer sleep quality. The total score ranges from 0 to 21.
Change in Major Depression Inventory | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Major Depression Inventory is a tool used to assess the severity of depression symptoms. It consists of a questionnaire with 10 items covering different aspects of depression, such as mood, sleep, appetite, and energy levels. Each item is rated on a scale from 0 to 5, with higher scores indicating more severe symptoms. The total score ranges from 0 to 50, with higher scores indicating a greater severity of depression.
Change in European Quality of life - 5 Dimensions | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The European Quality of Life-5 Dimensions is used to assess an individual's health-related quality of life. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels of severity: no problems, some problems, and extreme problems. The questionnaire provides a descriptive profile of an individual's health status based on their responses to these dimensions. The index score ranges from 0 to 1, where 1 represents full health and 0 represents a health state equivalent to death. Additionally, the EQ-5D includes a visual analog scale (VAS) where individuals rate their overall health on a scale from 0 to 100. This tool is widely used in health economics, clinical trials, and population health studies.
Change in Non-motor Symptoms Questionnaire | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Non-motor Symptoms Questionnaire is a 30-item questionnaire designed to assess the presence and severity of non-motor symptoms Parkinson's disease. The items of the NMSQuest are grouped to nine domains: gastrointestinal (8 items), urinary tract (2 items), sexual function (2 items), cardiovascular (2 items), apathy/attention/memory (3 items), hallucinations/delusions (2 items), depression/anxiety/anhedonia (2 items), sleep/fatigue (5 items), pain (1 item) and miscellaneous (3 items). For each item there is a yes or no answer.
Change in Brief Pain Inventory (Short Form) | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Brief Pain Inventory (Short Form) assesses pain severity and its impact on daily life. It asks about pain intensity, interference with activities, mood, and sleep. Additionally, it inquires about pain location and management strategies. Scores are calculated based on responses, with higher scores indicating more severe pain and greater interference with daily activities.
Change in The Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The MDS-UPDRS is a comprehensive assessment designed to monitor the burden and extent of Parkinson's disease. The MDS-UPDRS has 4 parts with a total summed score. Part I: non-motor experiences of daily living (13 questions). Part II: motor experiences of daily living (13 questions). Part III: motor examination (33 scores based on 18 questions with several right, left or other body distributions scores). Part IV: motor complications (6 questions). All items have 5 response options with uniform anchors of: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, 4 = severe). Higher scores indicate greater impact of PD symptoms.
Change in Six Minute Walk Test | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Six Minute Walk Test is a simple and widely used measure of functional exercise capacity. After the six minutes have elapsed, the total distance walked by the participant is recorded in meters. Longer distances indicate better functional exercise capacity and endurance.
Change in Timed Up and Go | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The participant is instructed to rise from a chair, walk a short distance (3 meters or 10 feet), turn around, walk back, and sit down again. The time taken to complete the task is recorded. Shorter time means better performance.
Change in Six Spot Step Test | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Six Spot Step Test is a functional assessment used to evaluate agility, coordination, and dynamic balance. The time taken to complete the sequence is recorded. Shorter time means better performance.
Change in Symbol Digit Modalities Test | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Symbol Digit Modalities Test is a cognitive assessment tool used to measure processing speed and attention. In this test, individuals are presented with a key that pairs symbols with numbers. The total score is based on the number of correct responses completed within a set time limit. A higher score indicates better cognitive function, reflecting faster processing speed and attention abilities.
Change in Montreal Cognitive Assessment | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The Montreal Cognitive Assessment is a widely used screening tool for detecting cognitive impairment. It evaluates various cognitive domains, including memory, attention, language, and visuospatial abilities. The test consists of tasks such as memory recall, naming, attention and concentration, abstraction, and orientation. Scores on the Montreal Cognitive Assessment range from 0 to 30, with higher scores indicating better cognitive function. A score of 26 or above is typically considered normal, although this may vary depending on factors such as age and education level.
Change in Muscle strength | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The dynamometer is used to measure muscle strength through maximal voluntary contractions. The patient will continue until a maximum has been found. Appropriate breaks are held between the repetitions.
Change in aerobic capacity | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  The VO2 max test measures the maximum amount of oxygen the patient can utilize during intense exercise. It involves wearing a face mask connected to a metabolic cart to analyze oxygen consumption and carbon dioxide production. The individual performs progressively intense exercise until reaching exhaustion while vital signs are monitored. The VO2 max is determined as the point at which oxygen consumption plateaus despite increasing exercise intensity. Higher VO2 max means better aerobic capacity = better health.
Change in Physical activity | Baseline, 12 weeks post test, 24 weeks follow up test, 36 weeks post test (resistance exercise group only)
  Patients are fitted with an accelerometer on their thigh and wear it for seven consecutive days. A higher score of counts per minute indicates greater physical activity, which corresponds to a better result.
Change in Rochester Fatigue Diary | 3. exercise session (week 2 in the intervention period) and 30. exercise session (week 12 in the intervention period). One answer every hour for 24 hours (excluding sleeping hours).
  The Rochester Fatigue Diary requires participants to rate their perceived level of fatigue every hour for 24 hours, beginning at 7 am, excluding sleeping hours. This fatigue diary will be answered two times during the intervention period. The rating is conducted using a Visual Analog Scale ranging from 0 to 100, where higher scores reflect greater fatigue.
Change in Visual Analog Scale for fatigue, tremor, bradykinesia, rigidity and postural instability | Monday, Wednesday and friday throughout the enrollment period (24 weeks for the aerobic exercise group and 36 weeks for the resistance exercise group)
  Fatigue, tremor, bradykinesia, rigidity and postural instability are scores on a Visual Analog Scale ranging from 0 to 100, where higher scores reflect greater impact of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Biology, Dep. of Public Health, Aarhus University, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langeskov-Christensen M, Hvid LG, Jensen HB, Nielsen HH, Petersen T, Stenager E, Dalgas U. Efficacy of high-intensity aerobic exercise on common multiple sclerosis symptoms. Acta Neurol Scand. 2022 Feb;145(2):229-238. doi: 10.1111/ane.13540. Epub 2021 Oct 22. PMID 34687036
- [Background] Riemenschneider M, Hvid LG, Ringgaard S, Nygaard MKE, Eskildsen SF, Petersen T, Stenager E, Dalgas U. Study protocol: randomised controlled trial evaluating exercise therapy as a supplemental treatment strategy in early multiple sclerosis: the Early Multiple Sclerosis Exercise Study (EMSES). BMJ Open. 2021 Jan 12;11(1):e043699. doi: 10.1136/bmjopen-2020-043699. PMID 33436475
- [Background] Riemenschneider M, Hvid LG, Ringgaard S, Nygaard MKE, Eskildsen SF, Gaemelke T, Magyari M, Jensen HB, Nielsen HH, Kant M, Falah M, Petersen T, Stenager E, Dalgas U. Investigating the potential disease-modifying and neuroprotective efficacy of exercise therapy early in the disease course of multiple sclerosis: The Early Multiple Sclerosis Exercise Study (EMSES). Mult Scler. 2022 Sep;28(10):1620-1629. doi: 10.1177/13524585221079200. Epub 2022 Mar 16. PMID 35296183
- [Background] Goetz CG, Poewe W, Rascol O, Sampaio C, Stebbins GT, Counsell C, Giladi N, Holloway RG, Moore CG, Wenning GK, Yahr MD, Seidl L; Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. Movement Disorder Society Task Force report on the Hoehn and Yahr staging scale: status and recommendations. Mov Disord. 2004 Sep;19(9):1020-8. doi: 10.1002/mds.20213. PMID 15372591
- [Background] Heine M, van de Port I, Rietberg MB, van Wegen EE, Kwakkel G. Exercise therapy for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2015 Sep 11;2015(9):CD009956. doi: 10.1002/14651858.CD009956.pub2. PMID 26358158
- [Background] Winward C, Sackley C, Meek C, Izadi H, Barker K, Wade D, Dawes H. Weekly exercise does not improve fatigue levels in Parkinson's disease. Mov Disord. 2012 Jan;27(1):143-6. doi: 10.1002/mds.23966. Epub 2011 Sep 27. PMID 21953509
- [Background] Rios Romenets S, Anang J, Fereshtehnejad SM, Pelletier A, Postuma R. Tango for treatment of motor and non-motor manifestations in Parkinson's disease: a randomized control study. Complement Ther Med. 2015 Apr;23(2):175-84. doi: 10.1016/j.ctim.2015.01.015. Epub 2015 Feb 9. PMID 25847555
- [Background] Solla P, Cugusi L, Bertoli M, Cereatti A, Della Croce U, Pani D, Fadda L, Cannas A, Marrosu F, Defazio G, Mercuro G. Sardinian Folk Dance for Individuals with Parkinson's Disease: A Randomized Controlled Pilot Trial. J Altern Complement Med. 2019 Mar;25(3):305-316. doi: 10.1089/acm.2018.0413. Epub 2019 Jan 9. PMID 30624952
- [Background] Shulman LM, Katzel LI, Ivey FM, Sorkin JD, Favors K, Anderson KE, Smith BA, Reich SG, Weiner WJ, Macko RF. Randomized clinical trial of 3 types of physical exercise for patients with Parkinson disease. JAMA Neurol. 2013 Feb;70(2):183-90. doi: 10.1001/jamaneurol.2013.646. PMID 23128427
- [Background] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037
- [Background] Granziera S, Alessandri A, Lazzaro A, Zara D, Scarpa A. Nordic Walking and Walking in Parkinson's disease: a randomized single-blind controlled trial. Aging Clin Exp Res. 2021 Apr;33(4):965-971. doi: 10.1007/s40520-020-01617-w. Epub 2020 Jun 11. PMID 32529596
- [Background] Atan T, Ozyemisci Taskiran O, Bora Tokcaer A, Kaymak Karatas G, Karakus Caliskan A, Karaoglan B. Effects of different percentages of body weight-supported treadmill training in Parkinson's disease: a double-blind randomized controlled trial. Turk J Med Sci. 2019 Aug 8;49(4):999-1007. doi: 10.3906/sag-1812-57. PMID 31292107
- [Background] Cugusi L, Solla P, Serpe R, Carzedda T, Piras L, Oggianu M, Gabba S, Di Blasio A, Bergamin M, Cannas A, Marrosu F, Mercuro G. Effects of a Nordic Walking program on motor and non-motor symptoms, functional performance and body composition in patients with Parkinson's disease. NeuroRehabilitation. 2015;37(2):245-54. doi: 10.3233/NRE-151257. PMID 26484516
- [Background] Ribas CG, Alves da Silva L, Correa MR, Teive HG, Valderramas S. Effectiveness of exergaming in improving functional balance, fatigue and quality of life in Parkinson's disease: A pilot randomized controlled trial. Parkinsonism Relat Disord. 2017 May;38:13-18. doi: 10.1016/j.parkreldis.2017.02.006. Epub 2017 Feb 7. PMID 28190675
- [Background] Dashtipour K, Johnson E, Kani C, Kani K, Hadi E, Ghamsary M, Pezeshkian S, Chen JJ. Effect of exercise on motor and nonmotor symptoms of Parkinson's disease. Parkinsons Dis. 2015;2015:586378. doi: 10.1155/2015/586378. Epub 2015 Feb 2. PMID 25722915
- [Background] Michels K, Dubaz O, Hornthal E, Bega D. "Dance Therapy" as a psychotherapeutic movement intervention in Parkinson's disease. Complement Ther Med. 2018 Oct;40:248-252. doi: 10.1016/j.ctim.2018.07.005. Epub 2018 Jul 7. PMID 30219460
- [Background] Herring MP, O'Connor PJ. The effect of acute resistance exercise on feelings of energy and fatigue. J Sports Sci. 2009 May;27(7):701-9. doi: 10.1080/02640410902777385. PMID 19424902
- [Background] Lin I, Edison B, Mantri S, Albert S, Daeschler M, Kopil C, Marras C, Chahine LM. Triggers and alleviating factors for fatigue in Parkinson's disease. PLoS One. 2021 Feb 4;16(2):e0245285. doi: 10.1371/journal.pone.0245285. eCollection 2021. PMID 33540422
- [Background] Alberts JL, Rosenfeldt AB. The Universal Prescription for Parkinson's Disease: Exercise. J Parkinsons Dis. 2020;10(s1):S21-S27. doi: 10.3233/JPD-202100. PMID 32925109
- [Background] Elbers RG, Verhoef J, van Wegen EE, Berendse HW, Kwakkel G. Interventions for fatigue in Parkinson's disease. Cochrane Database Syst Rev. 2015 Oct 8;2015(10):CD010925. doi: 10.1002/14651858.CD010925.pub2. PMID 26447539
- [Background] Siciliano M, Trojano L, Santangelo G, De Micco R, Tedeschi G, Tessitore A. Fatigue in Parkinson's disease: A systematic review and meta-analysis. Mov Disord. 2018 Nov;33(11):1712-1723. doi: 10.1002/mds.27461. Epub 2018 Sep 28. PMID 30264539
- [Background] Nassif DV, Pereira JS. Fatigue in Parkinson's disease: concepts and clinical approach. Psychogeriatrics. 2018 Mar;18(2):143-150. doi: 10.1111/psyg.12302. Epub 2018 Feb 6. PMID 29409156
- [Background] Port RJ, Rumsby M, Brown G, Harrison IF, Amjad A, Bale CJ. People with Parkinson's Disease: What Symptoms Do They Most Want to Improve and How Does This Change with Disease Duration? J Parkinsons Dis. 2021;11(2):715-724. doi: 10.3233/JPD-202346. PMID 33459664
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Tysnes OB, Storstein A. Epidemiology of Parkinson's disease. J Neural Transm (Vienna). 2017 Aug;124(8):901-905. doi: 10.1007/s00702-017-1686-y. Epub 2017 Feb 1. PMID 28150045